CLINICAL TRIAL: NCT05496140
Title: Remote School-Home Program to Improve Youth Attention and Behavior in Mexican Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLSRFUERTE 2; R21MH124066 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-12

CONDITIONS: ADHD; Oppositional Defiant Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Oppositional Defiant Disorder

STUDY DESIGN:
Intervention Model Description: 8-school clustered randomized controlled trial (RCT).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLS-R-FUERTE (Experimental): Active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  Interventions: Behavioral: CLS-R-FUERTE
- Care-As-Usual (No Intervention): Continued participation in school care-as-usual

INTERVENTIONS:
Behavioral: CLS-R-FUERTE — The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  Arms: CLS-R-FUERTE

SUMMARY:
Neurodevelopmental disorders of inattention and disruptive behavior, such as Attention-Deficit/ Hyperactivity Disorder (ADHD) and Oppositional Defiant Disorder (ODD), are among the most common youth mental health conditions across cultures. An efficacious and feasible solution to improving affected youth's ADHD/ODD is training existing school clinicians to deliver evidence-based intervention with fidelity. Despite initial promising results of training school clinicians to treat ADHD/ODD in settings suffering from high unmet need, such as Mexico, scalability is limited by a lack of researchers with capacity to train, monitor, and evaluate school clinicians in such efforts on a large scale. Thus, there is a need to develop more feasible interventions and training programs for school clinicians, as well as create a system with capacity for scalable training and evaluation, to combat the widespread impact ofADHD/ODD worldwide. Converting interventions and school clinician professional development programs for fully-remote delivery allows for more flexibility, accessibility, affordability, scalability, and promise for ongoing consultation than in-person options. Supporting scalable training for school clinicians could address a significant public health concern in Mexico, as only 14% of Mexican youth with mental health disorders receive treatment and less than half of those treated receive more than minimally adequate care. The study team is uniquely suited for this effort, given that they developed the only known school-home ADHD/ODD evidence-based intervention in Latin America-and-have developed a web-based training for U.S. school clinicians with promising preliminary results. The study team's prior studies and high levels of unmet need make Mexico an ideal location for this proposal; however, lessons learned could be used to expand scalable school clinician training for evidence-based intervention in other settings and/or for other disorders. Thus, this study focuses on comparing the fully-remote CLS-R-FUERTE program vs. care-as-usual in an 8-school clustered randomized controlled trial (RCT). The team predicts: 1) school clinicians trained in the remote program will be satisfied and show improved skills, 2) parents, youth, and teachers treated by school clinicians in the remote program will engage/adhere, and 3) youth in the remote program will show more ADHD/ODD improvements compared to care-as-usual

ELIGIBILITY:
Inclusion Criteria:

* Students meeting the following criteria are eligible:

  * at least six inattention symptoms and/or six hyperactive/impulsive symptoms endorsed by parent or teacher as occurring often or very often,
  * at least one area of impairment rated as concerning by both parent and teacher, and
  * a parent and teacher agreeing to participate.
  * Students taking medication are eligible as long as regimens were stable.
* Parents and teachers and school clinicians of participating are eligible to participate.

Exclusion Criteria:

All Participants: Anyone who does not speak and read Spanish will be excluded, given that all informed consent, measurement, and activity procedures will be conducted in Spanish.

Child Participants

* Children taking medication will be eligible for screening after the child has been on a stable medication regimen for at least one month (to minimize chance that treatment effects are due to medication and not the proposed program).
* Presence of conditions that are incompatible with this study's treatment.
* severe visual or hearing impairment,
* severe language delay,
* psychosis,
* Child does not read or speak Spanish (inability to complete assessment measures or participate in group treatments).
* Child is in an all-day special education classroom. Children in these classrooms are frequently receiving intensive behavior modification programs and assistance such that the teacher consultation component would be expected to require modification for use in these settings.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lauren M Haack, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Period: Overall Study
Arm/Group | CLS-R-FUERTE | Care-As-Usual
Started | 79; 4 Schools (This represents n = 27 students, n = 27 parents, n = 18 teachers and n = 7 school clinicians) | 84; 4 Schools (This represents n = 30 students, n = 30 parents, n = 19 teachers, and n = 5 school clinicians)
Completed | 79; 4 Schools (This represents n = 27 students, n = 27 parents, n = 18 teachers, and n = 7 school clinicians) | 84; 4 Schools (This represents n = 30 students, n = 30 parents, n = 19 teachers, and n = 5 school clinicians)
Not Completed | 0; 0 Schools | 0; 0 Schools

BASELINE CHARACTERISTICS:
Population: Total CLS-R-FUERTE N = 79
  Total Care-As-Usual N = 84
Groups:
- CLS-R-FUERTE -Students: Students active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  CLS-R-FUERTE: The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
- CLS-R-FUERTE -Parents: Parents active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  CLS-R-FUERTE: The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
- CLS-R-FUERTE -Teachers: Teachers active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  CLS-R-FUERTE: The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
- CLS-R-FUERTE -School Clinicians: School clinicians active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  CLS-R-FUERTE: The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
- Care-As-Usual - Students: Students continued participation in school care-as-usual
- Care-As-Usual - Parents: Parents continued participation in school care-as-usual
- Care-As-Usual - Teachers: Teachers continued participation in school care-as-usual
- Care-As-Usual - School Clinicians: School clinicians continued participation in school care-as-usual
- Total: Total of all reporting groups
Arm/Group | CLS-R-FUERTE -Students | CLS-R-FUERTE -Parents | CLS-R-FUERTE -Teachers | CLS-R-FUERTE -School Clinicians | Care-As-Usual - Students | Care-As-Usual - Parents | Care-As-Usual - Teachers | Care-As-Usual - School Clinicians | Total
Number analyzed (Participants) | 27 | 27 | 18 | 7 | 30 | 30 | 19 | 5 | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27 | 0 | 0 | 0 | 30 | 0 | 0 | 0 | 57
  Between 18 and 65 years | 0 | 27 | 18 | 7 | 0 | 30 | 19 | 5 | 106
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 27 | 18 | 6 | 11 | 30 | 16 | 4 | 116
  Male | 23 | 0 | 0 | 1 | 19 | 0 | 3 | 1 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 27 | 18 | 7 | 30 | 30 | 19 | 5 | 163
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Mexico | 27 | 27 | 18 | 7 | 30 | 30 | 19 | 5 | 163

OUTCOME MEASURES:

1. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Parent Checklist ADHD Combined Type Symptom Severity Score
Description: Parents will assess ADHD symptoms using the CSI-4. The CSI-4: Parent Checklist contains 18 symptoms for ADHD, Combined type (ADHD:C; 18 items). Each symptom is rated on a 4-point scale (0= never to 3= very often). The average of ADHD:C scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: The analysis solely focuses on the children cohort of the population, as the intervention is directed at children. Data were not analyzed for the adult population or any other cohort. As such, the Overall Number of Participants Analyzed represents only the children cohort.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: school
Groups:
- CLS-R-FUERTE - Students: Students active program participation in: a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). via school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
  CLS-R-FUERTE: The CLS-R-FUERTE program is a remote school clinician training and comprehensive psychosocial intervention designed to improve attention and behavior in Mexican school-aged youth (grades 1-5). It contains the same evidence-based service components to improve youth attention/behavior as the in-person CLS-FUERTE program; specifically, it features school clinician training by a clinical research team to lead parent skill groups, child skill groups, and teacher consultation in a behavioral classroom management system.
Arm/Group | CLS-R-FUERTE - Students | Care-As-Usual - Students
Number analyzed (Participants) | 27 | 30
Number analyzed (school) | 4 | 4
score on a scale
  Baseline | 1.73 (0.63) | 1.90 (0.60)
  Post treatment | 0.96 (0.51) | 1.43 (0.60)

2. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Teacher Checklist ADHD Combined Type Symptom Severity Score
Description: Teachers will assess ADHD symptoms using the CSI-4. The CSI-4: Teacher Checklist contains 18 symptoms for ADHD, Combined type (ADHD:C; 18 items). Each symptom is rated on a 4-point scale (0= never to 3= very often). The average of ADHD:C scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: school
Arm/Group | CLS-R-FUERTE - Students | Care-As-Usual - Students
Number analyzed (Participants) | 27 | 30
Number analyzed (school) | 4 | 4
score on a scale
  Baseline | 1.91 (0.63) | 1.81 (0.59)
  Post treatment | 1.20 (0.74) | 1.69 (0.60)

3. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Parent Checklist (Oppositional Defiant Disorder) ODD Symptom Severity Score
Description: Parents will assess ODD symptoms using the CSI-4. The CSI-4: Parent Checklist contains 9 symptoms of ODD. Each symptom is rated on a 4-point scale (0= never to 3= very often). The average ODD scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: school
Arm/Group | CLS-R-FUERTE - Students | Care-As-Usual - Students
Number analyzed (Participants) | 27 | 30
Number analyzed (school) | 4 | 4
score on a scale
  Baseline | 0.99 (0.63) | 1.31 (0.68)
  Post Treatment | 0.67 (0.47) | 1.10 (0.53)

4. Primary Outcome: Change in Child Symptom Inventory-4 (CSI-4) Teacher Checklist (Oppositional Defiant Disorder) ODD Symptom Severity Score
Description: Teachers will assess ODD symptoms using the CSI-4. The CSI-4: Teacher Checklist contains 9 symptoms of ODD. Each symptom is rated on a 4-point scale (0= never to 3= very often). The average ODD scores range from zero to four, with higher scores indicating more severe symptoms.
Time Frame: Baseline and post treatment (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: school
Arm/Group | CLS-R-FUERTE - Students | Care-As-Usual - Students
Number analyzed (Participants) | 27 | 30
Number analyzed (school) | 4 | 4
score on a scale
  Baseline | 1.19 (0.69) | 1.20 (0.90)
  Post Treatment | 0.88 (0.77) | 0.89 (0.86)

5. Primary Outcome: Change Impairment Rating Scale (IRS) Parent Questionnaire Overall Severity Score
Description: Parents will assess impairment using the IRS. The IRS Parent Questionnaire contains 8 items of functional impairment (i.e., academic and peer relations). Each item is rated on a 7-point scale (1= no problem; does not need treatment/services to 7= extreme impairment; definitely needs treatment/services). The average of all IRS scores range from one to seven, with higher scores indicating more severe impairment.
Time Frame: Baseline and post treatment (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: school
Arm/Group | CLS-R-FUERTE - Students | Care-As-Usual - Students
Number analyzed (Participants) | 27 | 30
Number analyzed (school) | 4 | 4
score on a scale
  Baseline | 4.03 (1.59) | 4.03 (1.33)
  Post treatment | 1.72 (0.80) | 2.36 (0.98)

6. Primary Outcome: Change Impairment Rating Scale (IRS) Teacher Questionnaire Overall Severity Score
Description: Teachers will assess impairment using the IRS. The IRS Teacher Questionnaire contains 8 items of functional impairment (i.e., academic and peer relations). Each item is rated on a 7-point scale (1= no problem; does not need treatment/services to 7= extreme impairment; definitely needs treatment/services). The average of all IRS scores range from one to seven, with higher scores indicating more severe impairment.
Time Frame: Baseline and post treatment (8 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: school
Arm/Group | CLS-R-FUERTE - Students | Care-As-Usual - Students
Number analyzed (Participants) | 27 | 30
Number analyzed (school) | 4 | 4
score on a scale
  Baseline | 5.01 (1.22) | 5.18 (1.08)
  Post treatment | 2.90 (1.51) | 3.59 (1.46)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 10 weeks.
Description: The total number of participants (N = 163) represents n = 57 students, n = 57 parents, n = 37 teachers and n = 12 school clinicians
Arm/Group | CLS-R-FUERTE | Care-As-Usual
All-Cause Mortality (participants affected / at risk) | 0/79 | 0/84
Serious Adverse Events (participants affected / at risk) | 0/79 | 0/84
Other Adverse Events (participants affected / at risk) | 0/79 | 0/84

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT05496140/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT05496140/ICF_001.pdf